CLINICAL TRIAL: NCT05756517
Title: Basic Mobility and Levels of Physical Activity During Hospitalization for a Hip Fracture: Functions Needed and Strategies Used
Brief Title: Basic Mobility and Physical Activity During Hospitalization for a Hip Fracture: Functions Needed and Strategies Used
Acronym: HIP-ME-UP
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Maria Swennergren Hansen, Post doc, Hvidovre University Hospital
Other Study IDs: HIP-ME-UP Study 1
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Present study aim to gain an understanding of functions needed and strategies used for patients following hip fracture surgery to be independent in basic mobility activities during acute hospitalization, and establish knowledge of how much (or little) patients get out of bed.

Within the patients included in this cohort study (1), a subgroup will also be included in a satellite study (2), with a separate objective. Definitions are presented in the detailed description below (objectives 1-2).

DETAILED DESCRIPTION:
The objectives are;

1. To determine levels of physical activity among a broad representation of patients hospitalized following hip fracture surgery, and secondly to explore the association with 30-day readmission, and mortality.
2. To understand and define which functions and strategies are needed for patients hospitalized following hip fracture surgery to be independent in the basic mobility activities: getting in/out of bed, sit-to-stand from a chair and walking.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone surgery for hip fracture at Hvidovre Hospital admitted to department 210/212 or at Bispebjerg Hospital department M1.
* Being able to participate in basic mobility activities with assistance pre-fracture (Cumulated Ambulation Score (by recall) ≥ 3)
* Able to give written informed consent or having a relative/legal guardian to give written consent, not later than on 3rd postoperative day

Exclusion Criteria:

* Postoperative weightbearing restrictions
* Multiple fractures
* Suspected pathological fracture due to cancer
* Terminal illness
* Post operative medical complications limiting the patient from getting out of bed
* Patients with permanent residence in a nursing home
* Patient unwilling to cooperate for testing

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Hvidovre Hospital and Bispebjerg Hospital. A subgroup of patients from Hvidovre Hospital will also be recruited to the basic mobility satelite study (being filmed on 3-5 post operative day). This subpoplulation has slight different eligibility criteria. Addition to the inclusion criteria below: their pre-fracture CAS =6, able to give written informed consent, not later than on 5th postoperative day and able to speak and understand Danish. Additional exclusion criteria: Post operative medical complications limiting the patient from participating in physio- or occupational therapy, history of stroke with motor disability, cognitive dysfunction determined by chart review, reported by nursing staff, or observed by trained research staff (disoriented, dementia, active delirium), patient unwilling to participate in rehabilitation post-operative or do not want to cooperate for testing and to be filmed during transfer out/in of bed
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Physical activity/upright time (time standing and walking) | Days of acute hospitalization (up to day 20)
  Will be measured using SENS Innovation Aps motion activity measurement system which is a waterproof activity sensor placed laterally on the right thigh.

SECONDARY OUTCOMES:
Basic mobility | Daily on weekdays during hospitalization (up to day 20)
  Will be measured using Cumulated Ambulation Score (CAS). The CAS score allows day-to-day measurements of basic mobility. It describes the patients' independence in three activities (getting in and out of bed, sit-to-stand from a chair, and walking), with each activity assessed on a three-point ordinal scale from 0 to 2, resulting in a total CAS between 0 and 6 (6 i maximum score indicating the patient to be independent in basic mobility).
Frailty | Registered at inclusion, but scored how they were 2 weeks before present hospitalization
  Will be assessed using Clinical Frailty Scale (CFS) which is a clinical judgement-based frailty tool. The CFS evaluates specific domains including comorbidity, function., and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
Cognitive status | At inclusion
  Will be assessed using the Short Orientation-Memory Concentration (OMC). It consists of a 6-item patient reported questionnaire and is validated as a measure of cognitive impairment. The score ranges from 0-28 where 0 is equal to normal cognition and 28 is appraised as a severe impairment.
Nutrition risk screening | At inclusion
  Will be assessed by using Mini Nutritional Assessment Short Form (MNA-SF) which is a validated tool often used within research in this field.It has 6 items and ranges from 0 (malnourished) to 14 (normal nutritional status).
Comorbidity | At inclusion
  Will be assessed using The American Society of Anesthesiologists (ASA) physical status classification system. The ASA score is a subjective assessment of a patient's overall health that is based on five classes. One means the patients is healthy and fit, and 5 is a moribund patient who is not expected to live 24 hour with or without surgery.
Pain at rest and walking | At inclusion, and at discharge (assessed up to day 20)
  Will be assessed using the 5-point Verbal Rating Scale (VRS, no pain, slight pain, moderate pain, severe pain, and unbearable pain) both at rest lying down and during walking.
Body strength | At inclusion and 3-5 days post-operative.
  Will be assessed using test of hand grip strength (HGS). Although the measure of HGS assesses the function of one muscle group, it is regarded as an indicator of overall body strength.
Pre-fracture physical activity | Registered at inclusion, but recall the last few weeks before present hospitalization
  Will be assessed using a validated questionnaire from the Swedish National Board of Health and Welfare, providing a total score from 3 to 19. A score ≥11 corresponds to fulfillment of the Word Health Organization's recommendation for weekly physical activity
Filming patients performing basic mobility activities | On the 3-5 post-operative day
  A subgroup of patients will be filmed when; (getting in and out of bed, sit-to-stand from a chair, and walking.
Data 30 days post discharge | 30 days post discharge
  Patient journal will be reviewed and there will be registered if the patient has been readmitted or has died.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Swennergren Hansen, PT, PhD, Principal Investigator — Department of Orthopedic Surgery and Department of Physio- and Occupational Therapy, Hvidovre Hospital
Locations (1):
- Department of Physio- and Occupational Therapy and Orthopedic Surgery, Copenhagen University Hospital, Amager-Hvidovre, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen MS, Wassar Kirk J, Kristensen MT, Kampp Zilmer C, Marie Skibdal K, Bandholm T, Pedersen MM; HIP-ME-UP Collaborative Group. Strategies used by patients when getting in and out of bed early after hip fracture surgery - The HIP-ME-UP cohort. Hosp Pract (1995). 2025 Feb;53(1):2491305. doi: 10.1080/21548331.2025.2491305. Epub 2025 Apr 30. PMID 40257221
- [Derived] Hansen MS, Kristensen MT, Zilmer CK, Berger AL, Kirk JW, Marie Skibdal K, Kallemose T, Bandholm T, Pedersen MM; HIP-ME-UP Collaborative Group. Very low levels of physical activity among patients hospitalized following hip fracture surgery: a prospective cohort study. Disabil Rehabil. 2025 Jan 21:1-10. doi: 10.1080/09638288.2025.2451769. Online ahead of print. PMID 39835691